CLINICAL TRIAL: NCT01270009
Title: Implication of the Antiapoptotic Protein BCL-B in the Pathogenesis of Multiple Myeloma
Brief Title: Role of BCL-B in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 09-PP-10
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
MM accounts for 10% of hematopoietic malignancies. Despite the use of various drug combinations in chemotherapy, life expectancy of MM patients does not exceed 7 years. Until now, lack of specific markers of the disease has not allowed efficient specific molecular targeting. In view of our preliminary results, the antiapoptotic protein Bcl-B could be a novel diagnostic and pronostic marker of MM. Therefore, our main objective will be to confirm that Bcl-B is indeed a novel diagnostic and pronostic marker and a new potential therapeutic target of MM. Targeting Bcl-2 family member's is a promising strategy for the treatment of hematopoietic malignancies. In this context, specific targeting of Bcl-B could improve the treatment of patients suffering MM. Of note, this could be achieved by converting the antiapoptotic function of Bcl-B to a proapoptotic one thanks to the use of small mimetic peptides derived from Nur77 one of its interactors.

ELIGIBILITY:
Patients with Multiple Myeloma and MGUS newly diagnosed at the Service de Medecine Interne-Cancerologie department of the Nice CHU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma and MGUS newly diagnosed at the Service de Medecine Interne-Cancerologie department of the Nice CHU
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine whether BCL-B is a survival factor in malignant plasmocytes, we will analyse the level of expression of Bcl-B at the both mRNA and protein levels in a cohort of MGUS and MM patients. | 6 months
  To determine whether BCL-B is a survival factor in malignant plasmocytes,we will analyse the level of expression of Bcl-B at the both mRNA and protein levels in a cohort of MGUS and MM patients. The implication of Bcl-B in malignant plasmocyte survival will be evaluated by loss of fucntion experiments (Si-RNA). This will also allow to determine whether Bcl-B is involved in the MGUS to MM transition.

SECONDARY OUTCOMES:
To determine whether deregulation of BCL-B expression is associated to chimioresistances commonly observed in Multiple Myeloma, We will compare Bcl-B expression in MM patients either sensitive or resistant to conventional therapies. | 6 months
  To determine whether deregulation of BCL-B expression is associated to chimioresistances commonly observed in Multiple Myeloma, We will compare Bcl-B expression in MM patients either sensitive or resistant to conventional therapies. We will focuse on resistance to Velcade. we have also isolated established MM cell lines resistant to velcade in vitro which will be useful for the study with MM patients samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Gabriel FUZIBET, MD, Principal Investigator — CHU de Nice Service de Médecine Interne et Cancérologie Hôpital de l'Archet
Locations (1):
- Service de Médecine interne et cancérologie - Hôpital de l'Archet, Nice, France